CLINICAL TRIAL: NCT01936389
Title: A Prospective Study to Assess the Hypotensive Efficacy of Rho-Kinase Inhibitor AR-12286 Ophthalmic Solution 0.5% and 0.7% in Patients With Exfoliation Syndrome and Ocular Hypertension or Glaucoma
Acronym: ROCK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robert Ritch, MD, LLC. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12286
Record Dates: First submitted 2013-08-28; First posted 2013-09-06 (Estimated); Results first posted 2015-04-24 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2015-04

CONDITIONS: Exfoliation Syndrome; Ocular Hypertension; Open Angle Glaucoma
MeSH Terms: conditions — Exfoliation Syndrome; Ocular Hypertension; Glaucoma, Open-Angle | interventions — AR-12286

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 0.5% (Experimental): 0.5% Rho-Kinase Inhibitor
  Interventions: Drug: AR-12286
- 0.7% (Experimental): 0.7% Rho-Kinase Inhibitor
  Interventions: Drug: AR-12286

INTERVENTIONS:
Drug: AR-12286
  Other Names: Rho-Kinase Inhibitor

SUMMARY:
Glaucoma is the world's the second leading cause of irreversible blindness. The World Health Organization (WHO) estimated the incidence of blindness due to glaucoma to be 4.4 million people worldwide in 2002. Intraocular pressure (IOP) is the sole proven modifiable risk factor for the development and progression of glaucomatous optic neuropathy. Medical therapy is aimed at lowering IOP in order to prevent or slow progression.

Exfoliation syndrome (XFS) is the most common identifiable cause of open-angle glaucoma, affecting an estimated 60 to 70 million people worldwide. Approximately two-thirds of patients have disease in only one eye on clinical examination; however, XFS is detectable in the other eye with conjunctival biopsy. XFS is also a systemic disease, with effects on the cardiovascular and cerebrovascular systems.

Patients with XFS are twice as likely to convert from ocular hypertension to glaucoma. Glaucoma in XFS is more severe than primary open angle glaucoma. There is greater diurnal IOP fluctuation, greater visual field loss and optic nerve head damage at the time of diagnosis, poorer response to medications, more rapid visual field progression and more frequent need for surgery.

Because you meet eligibility criteria for our study, we ask for your consent to participate in the study described below. In brief, you will be taking an investigational drug (AR-12286, rho-kinase Inhibitor) at either 0.5% or 0.7% once a day for 6 months. This drug is currently being tested in patients with primary open-angle glaucoma, but not yet in glaucoma in exfoliation syndrome. Because of the mechanism of glaucoma in XFS and the mechanism of action of rho-kinase inhibitors, there is reason to think it would be more effective in eyes with XFS and glaucoma than in primary open-angle glaucoma (ordinary glaucoma). There will be a baseline and study day 1 visit, week 1 visit, month 1 and 3 visit, week 13 visit, month 6 visit and a week 25 visit; for a total of 7 office visits.

ELIGIBILITY:
Inclusion Criteria:

* 50-85 y.o.
* Male and Female
* Exfoliation Syndrome and ocular hypertension or mild or moderate exfoliative glaucoma
* IOP ≥22 mmHg prior to initiation of treatment in one or both eyes with two measurements taken two hours apart
* No previous intraocular surgery except clear cornea phacoemulsification
* Corrected visual acuity in both eyes ≥20/50 in the eligible eye
* Not more than 6 diopters spherical equivalent on the study eye
* Not more than 3 diopters cylinder equivalent on the study eye
* Have given written informed consent, prior to any investigational procedures
* Ability to attend for the 6-month duration of the study

Exclusion Criteria:

* Open angle glaucoma other than exfoliative glaucoma
* Closed angle glaucoma (primary or secondary)
* Intraocular pressure >30 mm Hg
* Severe exfoliation glaucoma
* Known hypersensitivity to any component of the formulation (benzalkonium chloride, etc.), or to topical anesthetics
* Previous intraocular surgery except clear cornea phacoemulsification
* Clinically significant ocular disease (e.g. corneal edema, uveitis, severe keratoconjunctivitis sicca) which might interfere with the study
* Ocular medication of any kind within 30 days of base-line visit, with the exception of ocular hypotensive medications and/or lubricating drops for dry eye (which may be used throughout the study)
* Any abnormality preventing reliable applanation tonometry of either eye
* Clinically significant systemic disease (e.g., uncontrolled diabetes, myasthenia gravis, hepatic, renal, endocrine or cardiovascular disorders) which might interfere with the study
* Changes of systemic medication that could have a substantial effect on IOP anticipated during the study
* Participation in any investigational study within the past 30 days
* Inability to perform reliable VF testing
* Unwilling to sign the consent form approved by the Institutional Review Board (IRB) of the New York Eye and Ear Infirmary
* Self-reported poor compliance to treatment
* Reluctance to return for scheduled follow-up visits
* Patients not able to understand the nature of the study

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Glaucoma Associates of New York, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.5%: 0.5% Rho-Kinase Inhibitor
  AR-12286
- 0.7%: 0.7% Rho-Kinase Inhibitor
  AR-12286
Period: Overall Study
Arm/Group | 0.5% | 0.7%
Started | 5 | 5
Completed | 4 | 5
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5% | 0.7% | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 3 | 5 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Ocular Hypotensive Efficacy of Rho Kinase Inhibitor (AR-12286 0.5% and 0.7%)
Description: Goldmann Aplanation Tonometry (IOP mmHg) will be used to measure the ocular hypotensive efficacy.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 0.5% | 0.7%
Number analyzed (Participants) | 5 | 5
mmHg | 24.2 (2.4) | 25.8 (2.4)

ADVERSE EVENTS:
Arm/Group | 0.5% | 0.7%
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 1/5 | 0/5
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5% (N=5) | 0.7% (N=5)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No